CLINICAL TRIAL: NCT03030248
Title: Randomized Double Blind Controlled Trial for the Treatment of Nucleic Acid Amplification Test (NAAT)+/Toxin Enzyme Immunoassay (EIA)- Clostridium Difficile in the Hematology Oncology Population
Brief Title: Vancomycin for C Difficile NAAT+/EIA- Hematology Oncology Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Silvia Munoz-Price, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00028749
Record Dates: First submitted 2017-01-19; First posted 2017-01-24 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-07

CONDITIONS: Clostridium Difficile Infection; Hematologic Diseases; Bone Marrow Transplant; Oncologic Disorders
Keywords: microbiome; bone marrow transplantation; Clostridium difficile; metabolomics; vancomycin
MeSH Terms: conditions — Clostridium Infections; Hematologic Diseases | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups, one receiving oral vancomycin capsules, the other receiving oral placebo capsules.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The allocation status of patients within this study will be held in sealed envelopes by the unblinded research pharmacist on the team. Neither the main care provider, study physicians, or the patient will know of their group, until either the end of the study (after data analysis). We will also have a blinded pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vancomycin treated group (Active Comparator): This group will be given vancomycin oral capsules, 125 mg, every 6 hours, for 14 days.
  Interventions: Drug: Vancomycin Oral Capsule
- Placebo group (Placebo Comparator): This group will be given placebo oral capsules every 6 hours for 14 days.
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Vancomycin Oral Capsule — We have chosen oral vancomycin capsules as it is currently a standard of care for Clostridium difficile infections, is poorly absorbed by the intestines, and is easier to blind compared to oral vancomycin solution.
  Other Names: Vancocin hydrochloride Oral Capsule
  Arms: Vancomycin treated group
Drug: Placebo Oral Capsule — A capsule containing gelatin, polyethylene glycol, titanium dioxide, iron oxide, and FD&C blue No. 2. Contains the inactive ingredients of the vancomycin oral capsule, as mixed by the Froedtert Health Research Pharmacy.
  Arms: Placebo group

SUMMARY:
This study will randomized hematology oncology patients with active diarrhea and a NAAT positive/toxin EIA negative to either 14 days of oral vancomycin capsules or placebo. The study is designed to include 30 patients (15 per arm).

Outcomes will include C. difficile load using qPCR, VRE loads, structural and functional microbiome changes and frequency of bowel movements. All endpoints will be measured at several time points including days 0, 14, 21 and 90.

DETAILED DESCRIPTION:
The adverse health consequences resulting from antibiotic overtreatment of NAAT(+), toxin(-) patients may be particularly important in transplant recipients. The usual treatment prescribed for CDI at the Froedtert Memorial Lutheran Hospital is oral vancomycin. While this drug has excellent activity against C. difficile and commonly suppresses its growth to non-detection, it does not eradicate carriage and its use results in marked and prolonged disruption of the lower intestinal microbiota. Meanwhile, the degree of lower intestinal microbiota disruption at the time of HSCT engraftment has been demonstrated to be an independent predictor (controlling for other markers of underlying disease) of overall and transplant-related 3-year mortality.14 In addition, recent findings suggest that bone marrow suppressive effects of antibiotics, in this case potentially unnecessary oral vancomycin (which is not appreciably absorbed), may be solely mediated via microbiota disruption. All these data supports the notion that antibiotic treatment of NAAT(+), toxin(-) C. difficile patients might have significant negative repercussions without a clear clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hematology oncology inpatient units at Froedtert Memorial Lutheran Hospital
* New onset of diarrhea during hospitalization
* C. difficile clinical testing showing NAAT positive EIA negative results

Exclusion Criteria:

* Being unable to consent for self
* Inability to take enteral medications
* Unwillingness to enroll in study
* Patient has a documented allergy to vancomycin
* Patient has a documented life expectancy shorter than treatment course (14 days)
* Patient is unwilling or unable to provide stool samples in the outpatient setting after discharge
* Diagnosis of C. difficile colitis [NAAT (+) and toxin EIA (+) within 3 months of enrollment).
* New onset of abdominal distention within 24 hours prior to the onset of diarrhea during index admission
* Presence of toxic megacolon
* Presence of clinical sepsis. Sepsis will be defined as a Sequential [Sepsis-related] Organ Failure Assessment (SOFA) score of 2 points or more as per 2016 definitions
* Pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Clostridium difficile bacterial loads in the stool | Pre-treatment, 1, 7, 14, 21, 28, and 90 days past the beginning of treatment
  Changes in Clostridium difficile bacterial counts from stool as determined by quantitative polymerase chain reaction (PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Munoz-Price, M.D., Ph.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Participant data to be shared would consist of age categories, genders, treatment groups, Clostridium difficile status, microbiome profile and metabolic profile. The data will be anonymized to prevent the identification of individual patients from the data provided. The data would be made available through contacting the principal investigator directly.

REFERENCES:
- [Background] Lessa FC, Winston LG, McDonald LC; Emerging Infections Program C. difficile Surveillance Team. Burden of Clostridium difficile infection in the United States. N Engl J Med. 2015 Jun 11;372(24):2369-70. doi: 10.1056/NEJMc1505190. No abstract available. PMID 26061850
- [Background] Martin JS, Monaghan TM, Wilcox MH. Clostridium difficile infection: epidemiology, diagnosis and understanding transmission. Nat Rev Gastroenterol Hepatol. 2016 Apr;13(4):206-16. doi: 10.1038/nrgastro.2016.25. Epub 2016 Mar 9. PMID 26956066
- [Background] Theriot CM, Koenigsknecht MJ, Carlson PE Jr, Hatton GE, Nelson AM, Li B, Huffnagle GB, Z Li J, Young VB. Antibiotic-induced shifts in the mouse gut microbiome and metabolome increase susceptibility to Clostridium difficile infection. Nat Commun. 2014;5:3114. doi: 10.1038/ncomms4114. PMID 24445449
- [Background] Theriot CM, Bowman AA, Young VB. Antibiotic-Induced Alterations of the Gut Microbiota Alter Secondary Bile Acid Production and Allow for Clostridium difficile Spore Germination and Outgrowth in the Large Intestine. mSphere. 2016 Jan 6;1(1):e00045-15. doi: 10.1128/mSphere.00045-15. eCollection 2016 Jan-Feb. PMID 27239562
- [Background] Sethi AK, Al-Nassir WN, Nerandzic MM, Bobulsky GS, Donskey CJ. Persistence of skin contamination and environmental shedding of Clostridium difficile during and after treatment of C. difficile infection. Infect Control Hosp Epidemiol. 2010 Jan;31(1):21-7. doi: 10.1086/649016. PMID 19929371
- [Result] Aldrete SD, Kraft CS, Magee MJ, Chan A, Hutcherson D, Langston AA, Greenwell BI, Burd EM, Friedman-Moraco R. Risk factors and epidemiology of Clostridium difficile infection in hematopoietic stem cell transplant recipients during the peritransplant period. Transpl Infect Dis. 2017 Feb;19(1). doi: 10.1111/tid.12649. PMID 27943501
- [Result] Isaac S, Scher JU, Djukovic A, Jimenez N, Littman DR, Abramson SB, Pamer EG, Ubeda C. Short- and long-term effects of oral vancomycin on the human intestinal microbiota. J Antimicrob Chemother. 2017 Jan;72(1):128-136. doi: 10.1093/jac/dkw383. Epub 2016 Oct 5. PMID 27707993
- [Result] Polage CR, Gyorke CE, Kennedy MA, Leslie JL, Chin DL, Wang S, Nguyen HH, Huang B, Tang YW, Lee LW, Kim K, Taylor S, Romano PS, Panacek EA, Goodell PB, Solnick JV, Cohen SH. Overdiagnosis of Clostridium difficile Infection in the Molecular Test Era. JAMA Intern Med. 2015 Nov;175(11):1792-801. doi: 10.1001/jamainternmed.2015.4114. PMID 26348734